CLINICAL TRIAL: NCT06508632
Title: The Effect of Mandala Art Therapy (Coloring) on Nausea, Vomiting, Pain and Anxiety in Children Receiving Outpatient Chemotherapy
Brief Title: The Effect of Mandala on Nausea, Vomiting, Pain and Anxiety in Chemotherapy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Fahri AŞKAN, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: F ASKAN
Record Dates: First submitted 2024-07-08; First posted 2024-07-18 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Pain; Anxiety
Keywords: Mandala Art Therapy; Child; Nausea Vomiting; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental, randomised controlled, single-blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantal group (Experimental): Individual mandala activity will be carried out in all sample groups after admission to the clinic where they come to receive outpatient chemotherapy and when they start taking medication.
  Interventions: Behavioral: Mandala group
- Control Group (No Intervention): In this study, the control group will receive standard care.

INTERVENTIONS:
Behavioral: Mandala group — Individual mandala activity will be carried out in all sample groups after admission to the clinic where they come to receive outpatient chemotherapy and when they start taking medication. Children will color (paint).
  Other Names: Control group
  Arms: Experimantal group

SUMMARY:
To determine the effect of mandala art therapy (coloring) on nausea, vomiting, pain and anxiety in children receiving outpatient chemotherapy. The concept of cancer is used to describe a group of diseases that start from a single cell and show uncontrolled growth, proliferation and spread to surrounding tissues. The cooperation of the family and the healthcare team plays a major role in the success of the treatment. Surgical treatment, radiotherapy and chemotherapy are applied in its treatment. Art therapy, a method of distraction, is used to prevent pediatric oncology patients from focusing on the pain and stressful life events they experience. By having children do artistic activities in the hospital room, nurses can reduce symptom management, social isolation, and long-term negative social effects.

DETAILED DESCRIPTION:
Cancer treatment in children is determined according to the type of cancer, its stage and the child's general health condition. Treatment options include the following; chemotherapy, radiotherapy, surgery, immunotherapy and targeted therapy. The following problems are observed in children receiving chemotherapy in the short and long term: fever, fatigue, weight loss, pain, fatigue, anxiety, nausea and vomiting, changes in sleep and mood. 91% of oncology patients have benefited from Complementary and Alternative Medicine (CAM), such as art, to improve their general health, and painting, painting, music and dance, and mind-body therapies have been shown to have positive effects on the quality of life in pediatric oncology patients.

Art therapy in the pediatric oncology patient population. The American Art Therapy Association (AATA) (2013) defines art therapy as healing. Increasing the physical, mental and emotional well-being of individuals is considered as creative interventions of art production. These interventions have been widely used as alternative treatments for a variety of conditions, including cancer.

Although there is a significant amount of research on the effects of art therapies, there is a lack of research in the existing literature regarding their specific effects on symptoms such as nausea, vomiting, pain, and anxiety. However, the effects on quality of life are generally given more attention.

Among the art therapies; Mandala art therapy is a type of art therapy using circular patterns and symbols. In this therapy, participants explore their inner world and express their emotions by creating their own mandates. It gives individuals the opportunity to concretize the complex and abstract thoughts in their minds caused by their painful experiences. Emotions and thoughts are spontaneously embedded in artistic products such as sculpture, music, painting, marbling and mandala. Mandala therapy improves creativity and problem-solving skills by increasing emotional awareness and expression.

As a result, mandala art therapy can be used in the treatment of many different problems such as stress, anxiety, depression, trauma and chronic disease, as well as in the management of symptoms.

To determine the sample size of the study, the power of the study was calculated with the G-Power 3.1.9.2 program using the confidence interval and effect size parameters. 80% power, 95% confidence interval and effect size of 0.5 or more. In the G-Power 3.1.9.2 program, the total sample size was calculated as 48 (24+24) based on 0.05 significance, 0.80 large effect and 80% power. However, considering the 10% loss and taking into account the parametric test assumption, the sample number of each group was determined as 30 people in the intervention group and 30 people in the control group, for a total of 60 people.

ELIGIBILITY:
Inclusion Criteria:

* Being at the pediatric chemotherapy clinic to receive outpatient chemotherapy
* Receiving daily chemotherapy
* Those who agreed to participate in the research
* Mother and child must know Turkish
* The child knows colors

Exclusion Criteria:

* Having a mental health problem (preventing the use of Mandala therapy coloring technique)
* Having a disability that prevents you from seeing or using your hand (a condition that prevents you from using the Mandala therapy coloring technique)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Rating scale | Approximately 2 hours from start
  It is a visual analog scale used to evaluate the intensity of pain. This scale includes six different facial expressions scored from 0 to 10. 0 means "no pain," while 10 means "most severe pain." The scale is used to diagnose pain in children aged 3-18. Pain scores are given according to the numerical values given to the faces on the scale. The lowest score is "1" and the highest score is "5". As the score from the scale increases, pain tolerance decreases, and as the score decreases, tolerance increases.

SECONDARY OUTCOMES:
Nausea and Vomiting Thermometer in Children with Cancer | Approximately 2 hours from start
  The Nausea and Vomiting Thermometer Scale in Children with Cancer is a tool used to evaluate the frequency and severity of nausea and vomiting in children with cancer aged 0-18 years. The structure of the scale consists of 2 subscales: Nausea: 0 (no nausea) - 10 (most severe nausea), Vomiting: 0 (no vomiting) - 10 (most severe vomiting), Visuals using 5 different colors and emojis for each subscale. A thermometer was created.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova University Balcalı Training and Research Hospital, Adana, Balçalı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided